CLINICAL TRIAL: NCT00144690
Title: A Double-Blind, Placebo-Controlled, Dose-Escalation, Parallel-Group Study of E2007 Given as Adjunctive Therapy in Patients With Refractory Partial Seizures
Brief Title: E2007 Given as Adjunctive Therapy in Patients With Refractory Partial Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-A001-206; 2005-004199-18 (EudraCT Number)
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Epilepsy
Keywords: Epilepsy refractory partial seizures
MeSH Terms: conditions — Epilepsy | interventions — perampanel

INTERVENTIONS:
Drug: E2007 (perampanel)
Drug: Placebo

SUMMARY:
The primary objective of this study is to determine the maximal tolerated dose (MTD) of E2007 given twice daily (bid) or once a day (qd) in patients with refractory partial-onset seizures (including secondarily generalized seizures). The secondary objectives are to evaluate the safety, efficacy, concentration-efficacy relationship, and pharmacokinetics of E2007 and the effects of E2007 on the Profile of Mood States (POMS) test.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent signed by patient or legal guardian prior to entering the study or undergoing any study procedures.
* Are reliable and willing to make themselves available for the study period and are able to record seizures and report adverse events themselves or have a caregiver who can record and report the events.
* Male and female patients will be eligible for enrollment. Females should be either of non-childbearing potential as a result of surgery, radiational therapy, menopause (one year post onset), or of childbearing potential and practicing a medically acceptable method of contraception (eg, abstinence, a barrier method plus spermicide, or intrauterine device [IUD]) for at least three months before Visit 1 (Screening) and for two months after the end of the study. They must also have a negative serum beta-human chorionic gonadotropin (beta-hCG) at Screening. Pregnant and/or lactating females are excluded. Those women using an oral contraceptive must also be using an additional approved method of contraception (eg, a barrier method plus spermicide, or IUD) starting with the Baseline Phase and continuing throughout the entire study period.
* Are between the ages of 18 and 70 years of age, inclusive.
* Are of 40 kg (88 lb) of weight or more.
* Have the diagnosis of epilepsy with partial-onset seizures with or without secondarily generalized seizures according to the International League Against Epilepsy's Classification of Epileptic Seizures (1981). Diagnosis should have been established by clinical history, electroencephalogram (EEG) and computed tomography/magnetic resonance imaging (CT/MRI) of the brain performed within the last 10 years and consistent with localization-related epilepsy.
* Have uncontrolled partial seizures despite having been treated with at least three different anti-epileptic drugs (AEDs) (given concurrently or sequentially) for at least 2 years.
* To be enrolled, patient must have averaged at least 4 partial seizures per month, with no 21-day seizure-free period during the 2 months preceding randomization. To be randomized, the patient must have had at least 3 seizures during the prospective Baseline Phase (28 days), with no 21-day seizure-free period. This should be documented in the form of medical history, medical records, or photocopied records of the patient diary/patient chart. Simple partial seizures without motor signs will not be counted towards this inclusion criterion.
* Are currently being treated with one or a maximum of two licensed AEDs and are known to take their medication(s) as directed.
* Are on a stable dose(s) of the same AED(s) for the 2 months prior to Visit 1.
* If using a vagal nerve stimulator, it must have been implanted for at least 5 months prior to Visit 1. Stimulator parameters may not be changed for at least 1 month prior to Visit 1 or thereafter during the study. Magnet use will be allowed and documented throughout the study.

Exclusion Criteria:

* Have participated in a study involving administration of an investigational compound within one month of Visit 1 (Screening), or within 5 half-lives of the previous investigational compound, whichever is longer.
* Presence of non-motor simple partial seizures only.
* Presence of primary generalized epilepsies or seizures, such as absences, myoclonic epilepsies, Lennox-Gastaut syndrome.
* History of status epilepticus in the past year or seizure clusters where individual seizures cannot be counted.
* Show evidence of clinically significant disease (cardiac, respiratory, gastrointestinal, renal disease, etc) that in the opinion of the Investigator(s) could affect the patient's safety or trial conduct.
* Show evidence of significant active hepatic disease. Stable elevations of liver enzymes, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) due to concomitant medication(s) will be allowed if they are less than 2 times the upper limit of normal (ULN).
* Show evidence of significant active hematological disease. White blood cell (WBC) count cannot be <= 2500/µL or an absolute neutrophil count <= 1000/µL.
* Clinically significant electrocardiogram (ECG) abnormality, including prolonged QTc defined as >= 450 msec for males and >= 470 msec for females.
* Presence of major active psychiatric disease. Patients taking a stable dose of selective serotonin reuptake inhibitor (SSRI) antidepressant will be allowed (except fluvoxamine).
* Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and tumors.
* Have a history of psychogenic seizures.
* Have a history of drug abuse and/or positive finding on urinary drug screening, other than prescribed medication.
* Have a history of alcohol abuse in the past 2 years, and/or positive finding on urinary drug screen.
* Have had multiple drug allergies (dermatological, hematological or organ toxicity) or one or more severe drug reactions.
* Allergy to lactose.
* Concomitant use of felbamate or use of felbamate within 2 months prior to Visit 1.
* Concomitant use of vigabatrin. Patients that took vigabatrin in the past must be off vigabatrin for at least 5 months prior to Visit 1 and must not have evidence of a clinically significant abnormality in a visual perimetry test.
* Concomitant use or use within the previous 4 weeks prior to Visit 1 of neuroleptics, monoamine oxidase (MAO) inhibitors, barbiturates (except for seizure control indication), benzodiazepines (other than occasional intermittent use), and narcotic analgesics.
* Frequent need of rescue benzodiazepines (one or more times a month).

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of E2007 given bid or qd in patients with refractory partial-onset seizures (including secondarily generalized seizures)

SECONDARY OUTCOMES:
To evaluate the safety, efficacy, and concentration-efficacy relationship

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Arroyo, M.D., Ph.D., Study Director — Eisai Inc.
Locations (5):
- United States (5):
  - Dept. of Neuro Surgery, Little Rock, Arkansas
  - USF Physicians Group, Tampa, Florida
  - Clinical Trials, Detroit, Michigan
  - Medical College of Ohio Comprehensive Epilepsy Ctr., Toledo, Ohio
  - Vanderbilt University Medical Ctr., Nashville, Tennessee

REFERENCES:
- [Result] Krauss GL, Bar M, Biton V, Klapper JA, Rektor I, Vaiciene-Magistris N, Squillacote D, Kumar D. Tolerability and safety of perampanel: two randomized dose-escalation studies. Acta Neurol Scand. 2012 Jan;125(1):8-15. doi: 10.1111/j.1600-0404.2011.01588.x. Epub 2011 Aug 29. PMID 21883097
- [Derived] Bresnahan R, Hill RA, Wang J. Perampanel add-on for drug-resistant focal epilepsy. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD010961. doi: 10.1002/14651858.CD010961.pub2. PMID 37059702
- [Derived] Maguire M. Response to "Perampanel and pregnancy: Could experience be a gloomy lantern that does not even illuminate its bearer?". Epilepsy Behav. 2022 Apr;129:108654. doi: 10.1016/j.yebeh.2022.108654. Epub 2022 Mar 16. No abstract available. PMID 35305920